CLINICAL TRIAL: NCT02049320
Title: Remifentanil for Sedation of Patients With Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman - Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00478
Record Dates: First submitted 2014-01-13; First posted 2014-01-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Remifentanil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remifentanil: Patients sedated using Remifentanil
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil

SUMMARY:
This is a descriptive retrospective study designed to measure the efficacy of remifentanil sedation and the ability to perform frequent neurological examinations of patients with traumatic brain injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously admitted to the hospital presenting with traumatic brain injury (TBI)
* Patients who have undergone sedation after presenting with TBI

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering a traumatic brain injury who were sedated in the PICU using remifentanil.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Depth of Sedation | Every 24 hrs until discharged from the PICU, up to 1 month.
  Sedation scores will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States